CLINICAL TRIAL: NCT00504842
Title: A Phase 1-2, Randomized, Placebo-Controlled, Single-Blind, Dose Escalation Study to Evaluate the Safety, Tolerability, and Activity of Ascending Single Doses of MRX-801 With Continuous Ultrasound Administration in Subjects With Acute Ischemic Stroke Receiving Treatment With Intravenous Tissue Plasminogen Activator
Brief Title: Transcranial Ultrasound in Clinical SONothrombolysis
Acronym: TUCSON
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: ImaRx Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRX-06-101-CP-01-01
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Microbubbles; Transcranial Doppler ultrasound; TIBI; Symptomatic Intracranial Hemorrhage; modified Rankin Scale; Recanalization; Perflutren
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: MRX-801
Drug: Placebo

SUMMARY:
This is a randomized, placebo controlled, parallel group dose escalation trial to evaluate the safety, tolerability, and activity of four sequential dose tiers of MRX-801 and ultrasound as an adjunctive therapy to tissue plasminogen activator (tPA) treatment in subjects with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Occlusion demonstrated by transcranial Doppler ultrasound
* Eligible for tPA

Exclusion Criteria:

* Right to left cardiac shunt
* Moderate to severe COPD
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-12; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic intracranial hemorrhage | 36 hours

SECONDARY OUTCOMES:
Rate of recanalization of occluded artery | 120 minutes
Independent outcome (modified Rankin Scale 0-2) | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Molina Cateriano, MD, Study Director — University Hospital Vall d'Hebron, Barcelona, Spain
Locations (14):
- United States (13):
  - University of Alabama, Birmingham, Alabama
  - Barrow Neurology Clinics at St. Joseph's Hospital, Phoenix, Arizona
  - Hoag Memorial Hospital, Newport Beach, California
  - California Pacific Medical Center, San Francisco, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Christiana Care Health System, Newark, Delaware
  - University of Miami, Miami, Florida
  - St. Louis University School of Medicine, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Methodist Hospital Neurological Institute, Houston, Texas
  - University of Texas, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
- Bichat - Claude Bernard University Hospital and Medical School, Paris, France